CLINICAL TRIAL: NCT01181050
Title: A Randomised, Single-dose, Double-blind, Placebo-controlled, Parallel-group Trial to Assess Clinical Efficacy of NNC0142-0002 in Subjects With Active Rheumatoid Arthritis
Brief Title: Efficacy of NNC0142-0002 in Subjects With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8555-3796; U1111-1114-9194 (Other: WHO); 2010-019261-28 (EudraCT Number)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid | interventions — NNC0142-0002 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4.0 mg/kg (Experimental): Subjects received a single dose of 4 mg/kg NNC0142-0002
  Interventions: Drug: NNC0142-0002
- Placebo (Placebo Comparator): Subjects received a single dose of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0142-0002 — A single dose of 4 mg NNC 0142-0000-0002/kg bodyweight. Administered subcutaneously (s.c., under the skin).
  Arms: 4.0 mg/kg
Drug: placebo — A single dose of 4 mg NNC 0142-0000-0002 placebo/kg bodyweight. Administered subcutaneously (s.c., under the skin).
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the clinical efficacy of a single dose of NNC0142-0002 administered to subjects with active rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of RA meeting the American College of Rheumatology 1987 (ACR1987) criteria, obtained at least three months prior to dosing with the trial product
* Subjects with active RA having a Disease Activity Score (DAS28-CRP) of 4.5 or more, at least five tender and five swollen joints (can be the same), including one swollen wrist or at least two swollen ipsilateral metacarpophalangeal (MCP) joints (second to fifth)
* Concomitant treatment with methotrexate (MTX) (7.5-25 mg/week) for at least 12 weeks, with stable dose for at least 4 weeks prior to dosing
* Ability to be examined by Magnetic Resonance Imaging (MRI)
* Having failed no biologic therapies for RA and no more than two non-biologic disease modifying antirheumatic drugs

Exclusion Criteria:

* Chronic inflammatory autoimmune disease other than RA (rheumatoid arthritis)
* Any ongoing chronic or active infectious disease or microbial infection requiring systemic oral or intravenous treatment against infection within 1 month prior to trial start
* Body mass index (BMI) below or equal to 18 or above or equal to 40 kg/m^2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Berlin, Germany
- Moscow, Russia
- Kiev, Ukraine

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 8 trial sites in 3 different countries (Germany, the Russian Federation and Ukraine) as follows: Germany: 1 site, the Russian Federation: 6 sites and Ukraine: 1 site. All sites enrolled, randomised and dosed at least 1 subject.
Period: Overall Study
Arm/Group | 4.0 mg/kg | Placebo
Started | 41 | 22
Completed | 41 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4.0 mg/kg | Placebo | Total
Number analyzed (Participants) | 41 | 22 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (10.8) | 52.0 (10.8) | 52.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 19 | 57
  Male | 3 | 3 | 6
DAS28-CRP (Disease Activity Score based on count of 28 joints and the C-reactive protein) [Mean (Standard Deviation); unit: scores] — DAS28-CRP=0.56×sqrt(tender joints [count:1-28])+0.28×sqrt(swollen joints [count:1-28])+0.36×Ln(CRP level+1)+0.014×(patient's disease assessment on 0-100 mm scale [100=most severe])+0.96. Range: 0.96 to no upper limit. Higher score=more severe disease
  scores | 5.4 (0.9) | 5.4 (1.0) | 5.4 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in DAS28-CRP After 12 Weeks of Treatment
Description: DAS28-CRP=0.56×sqrt(tender joints [count:1-28])+0.28×sqrt(swollen joints [count:1-28])+0.36×Ln(CRP level+1)+0.014×(patient's disease assessment on 0-100 mm scale [100=most severe])+0.96. Range: 0.96 to no upper limit. Higher score=more severe disease. Mean change in DAS-CRP score after 12 Weeks of treatment.
Time Frame: Week 0, Week 12
Population: Change in DAS28-CRP was calculated by using last observation carried forward method.
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | 4.0 mg/kg | Placebo
Number analyzed (Participants) | 41 | 22
scores | -1.0 (1.0) | -1.0 (1.0)
Statistical Analysis 1: Comparison: 4.0 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.9334, Mixed effect model repeated measures; Treatment difference = -0.02, 95% CI [-0.54 to 0.50]

2. Secondary Outcome: Change in DAS28-CRP After 6 Weeks of Treatment.
Description: DAS28-CRP=0.56×sqrt(tender joints [count:1-28])+0.28×sqrt(swollen joints [count:1-28])+0.36×Ln(CRP level+1)+0.014×(patient's disease assessment on 0-100 mm scale [100=most severe])+0.96. Range: 0.96 to no upper limit. Higher score=more severe disease. Mean change in DAS-CRP score after 6 Weeks of treatment.
Time Frame: Week 0, Week 6
Population: Change in DAS28-CRP was calculated by using last observation carried forward method.
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | 4.0 mg/kg | Placebo
Number analyzed (Participants) | 41 | 22
scores | -0.9 (1.1) | -1.0 (0.8)
Statistical Analysis 1: Comparison: 4.0 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.8293, Mixed effect model repeated measures; Treatment difference = 0.06, 95% CI [-0.46 to 0.58]

3. Secondary Outcome: Change in DAS28-CRP After 24 Weeks of Treatment.
Description: DAS28-CRP=0.56×sqrt(tender joints [count:1-28])+0.28×sqrt(swollen joints [count:1-28])+0.36×Ln(CRP level+1)+0.014×(patient's disease assessment on 0-100 mm scale [100=most severe])+0.96. Range: 0.96 to no upper limit. Higher score=more severe disease. Mean change in DAS-CRP score after 24 Weeks of treatment.
Time Frame: Week 0, Week 24
Population: Change in DAS28-CRP was calculated by using last observation carried forward method.
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | 4.0 mg/kg | Placebo
Number analyzed (Participants) | 41 | 22
scores | -1.3 (1.1) | -1.3 (1.1)
Statistical Analysis 1: Comparison: 4.0 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.8867, Mixed effect model repeated measures; Treatment difference = -0.04, 95% CI [-0.65 to 0.56]

ADVERSE EVENTS:
Time Frame: The adverse events were collected from dosing until end of trial (a total of 24 weeks)
Description: Safety analysis set includes all subjects who received one dose of the investigational product or its comparator
Arm/Group | 4.0 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/41 | 1/22
Other Adverse Events (participants affected / at risk) | 5/41 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4.0 mg/kg (N=41) | Placebo (N=22)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4.0 mg/kg (N=41) | Placebo (N=22)
Respiratory tract infection viral (Infections and infestations) | 1 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
As per protocol, this clinical proof-of-principle trial investigated a limited number of participants and doses (single-dose regimen).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to defer data release until specified milestones, e.g. availability of a clinical trial report. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property. Novo Nordisk reserves the right to prior review of site-specific publications and to ask for deferment of publication of individual site results until after the primary manuscript is accepted for publication.